CLINICAL TRIAL: NCT00730626
Title: Dose Response Study of the Impact of a Yogurt Containing Bifidobacterium Lactis BB-12 and Lactobacillus Acidophilus LA-5 on the Immune System and Gut Health.
Brief Title: Dose Response Study of a Fermented Yogurt on the Immune System and Gut Health
Acronym: PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Aliments ULTIMA Foods Inc. (Industry); McGill University (Other); TransBiothec (Unknown)
Responsible Party: Benoît Lamarche, Study Principal Investigator, Institute of Nutraceuticals and Functional Foods (INAF), Laval University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: INAF-119
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Immune System
Keywords: Probiotics; Immunity; Immune response; Intestinal microflora; Blood lipids; Phagocytosis activity
MeSH Terms: interventions — Yogurt

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): L.acidophilus and B.lactis (1x10E9 of each probiotics) with 40 mg of green the extract
  Interventions: Dietary Supplement: Yogurt with 1X10E9 BB-12 and LA-5
- 2 (Experimental): L.acidophilus and B.lactis (1x 10E10 of each probiotics) with 40 mg of green tea extract
  Interventions: Dietary Supplement: Yogurt with 1X10E10 BB-12 and LA-5
- 3 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Yogurt Placebo

INTERVENTIONS:
Dietary Supplement: Yogurt with 1X10E9 BB-12 and LA-5 — 100g of yogurt containing the probiotics L.acidophilus and B.lactis (concentrations of 1x10E9 of each probiotics) with 40 mg of green tea extract, once a day for 10 weeks.
  Arms: 1
Dietary Supplement: Yogurt with 1X10E10 BB-12 and LA-5 — 100g of yogurt containing the probiotics L.acidophilus and B.lactis (concentrations of 1x10E10 of each probiotics) with 40 mg of green tea extract, once a day for 10 weeks.
  Arms: 2
Dietary Supplement: Yogurt Placebo — 100g of yogurt placebo containing no probiotics and no green tea extract, once a day for 10 weeks.
  Arms: 3

SUMMARY:
The purpose of this study is to determine the dose-response effect of a yogurt containing a combination of bifidobacterium Lactis (BB-12) and Lactobacillus Acidophilus (LA-5) and green tea extract on markers of the immune system and gut health in healthy subjects. We hypothesize that the response of the immune function will be dose-dependent of the probiotics found in the fermented yogurt.

DETAILED DESCRIPTION:
There is an increasing list of food containing probiotics on the market. Several studies have emphasized the health benefits of single probiotics, particularly on the immune system. However, it is unclear how a combination of two different probiotics complemented with green tea extract can beneficially modify markers of the immune.

The aim of this study is to determine the dose-response effect of a yogurt containing a combination of bifidobacterium lactis (BB-12) and Lactobacillus Acidophilus LA-5 and green tea extract on immune system in healthy subjects. More specifically, this randomized, parallel placebo controlled study will investigate the impact of increasing doses (109 and 1010) of these probiotics on phagocytosis activity, oxidative metabolism and on the antipneumococcics antibody specific serotype response S. pneumoniae vaccination. Finally, this study will also examine the effect of increasing dose of these probiotics on intestinal microflora and blood lipids.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 55 years
* Healthy individuals, non-smokers
* BMI between 18 and 35 kg/m2
* Stable weight (+/- 5kg) for 3 months before randomisation
* Agree to receive a vaccine Pneumovax 23®

Exclusion Criteria:

* Pregnant or lactating woman
* Previous history of cardiovascular disease
* Diabetes
* Kidney or liver disease
* Gastrointestinal disorders or diseases
* Endocrine disorders or diseases
* Allergy
* Subjects taking hypolipidemic drugs, antidepressant, medication for high blood pressure, for inflammation or auto-immune diseases.
* Subject who have receive antipneumococcics vaccine in the year before randomisation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Phagocytosis activity and oxidative metabolism in phagocytes. | 6 weeks after vaccination

SECONDARY OUTCOMES:
antipneumococcics antibody specific serotype response to S. pneumoniae vaccination. | 6 weeks after yogurt consumption and vaccination
Intestinal microflora characteristics. | 4 weeks after yogurt consumption
Influence of blood lipids. | After 4 weeks and 10 weeks of yogurt consumption

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Lamarche, PhD, Principal Investigator — Institute of Nutraceuticals and Functional Foods (INAF), Laval University.; Jacques Hébert, MD, Study Director — Faculty of Medicine, Laval University.
Locations (1):
- Institute of Nutraceuticals and Functional Foods (INAF), Laval University, Québec, Quebec, Canada

REFERENCES:
- [Background] Winkler P, de Vrese M, Laue Ch, Schrezenmeir J. Effect of a dietary supplement containing probiotic bacteria plus vitamins and minerals on common cold infections and cellular immune parameters. Int J Clin Pharmacol Ther. 2005 Jul;43(7):318-26. doi: 10.5414/cpp43318. PMID 16035374
- [Background] de Vrese M, Winkler P, Rautenberg P, Harder T, Noah C, Laue C, Ott S, Hampe J, Schreiber S, Heller K, Schrezenmeir J. Probiotic bacteria reduced duration and severity but not the incidence of common cold episodes in a double blind, randomized, controlled trial. Vaccine. 2006 Nov 10;24(44-46):6670-4. doi: 10.1016/j.vaccine.2006.05.048. Epub 2006 Jun 6. PMID 16844267
- [Background] Kukkonen K, Nieminen T, Poussa T, Savilahti E, Kuitunen M. Effect of probiotics on vaccine antibody responses in infancy--a randomized placebo-controlled double-blind trial. Pediatr Allergy Immunol. 2006 Sep;17(6):416-21. doi: 10.1111/j.1399-3038.2006.00420.x. PMID 16925686
- [Background] Taylor AL, Hale J, Wiltschut J, Lehmann H, Dunstan JA, Prescott SL. Effects of probiotic supplementation for the first 6 months of life on allergen- and vaccine-specific immune responses. Clin Exp Allergy. 2006 Oct;36(10):1227-35. doi: 10.1111/j.1365-2222.2006.02553.x. PMID 17014429
- [Background] Olivares M, Diaz-Ropero MP, Sierra S, Lara-Villoslada F, Fonolla J, Navas M, Rodriguez JM, Xaus J. Oral intake of Lactobacillus fermentum CECT5716 enhances the effects of influenza vaccination. Nutrition. 2007 Mar;23(3):254-60. doi: 10.1016/j.nut.2007.01.004. PMID 17352961
- [Background] Schiffrin EJ, Brassart D, Servin AL, Rochat F, Donnet-Hughes A. Immune modulation of blood leukocytes in humans by lactic acid bacteria: criteria for strain selection. Am J Clin Nutr. 1997 Aug;66(2):515S-520S. doi: 10.1093/ajcn/66.2.515S. PMID 9250141
- [Background] Arunachalam K, Gill HS, Chandra RK. Enhancement of natural immune function by dietary consumption of Bifidobacterium lactis (HN019). Eur J Clin Nutr. 2000 Mar;54(3):263-7. doi: 10.1038/sj.ejcn.1600938. PMID 10713750
- [Background] Gill HS, Rutherfurd KJ, Cross ML, Gopal PK. Enhancement of immunity in the elderly by dietary supplementation with the probiotic Bifidobacterium lactis HN019. Am J Clin Nutr. 2001 Dec;74(6):833-9. doi: 10.1093/ajcn/74.6.833. PMID 11722966
- [Background] Roller M, Clune Y, Collins K, Rechkemmer G, Watzl B. Consumption of prebiotic inulin enriched with oligofructose in combination with the probiotics Lactobacillus rhamnosus and Bifidobacterium lactis has minor effects on selected immune parameters in polypectomised and colon cancer patients. Br J Nutr. 2007 Apr;97(4):676-84. doi: 10.1017/S0007114507450292. PMID 17349080
- [Background] Olivares M, Diaz-Ropero MP, Gomez N, Lara-Villoslada F, Sierra S, Maldonado JA, Martin R, Rodriguez JM, Xaus J. The consumption of two new probiotic strains, Lactobacillus gasseri CECT 5714 and Lactobacillus coryniformis CECT 5711, boosts the immune system of healthy humans. Int Microbiol. 2006 Mar;9(1):47-52. PMID 16636989
- [Derived] Savard P, Lamarche B, Paradis ME, Thiboutot H, Laurin E, Roy D. Impact of Bifidobacterium animalis subsp. lactis BB-12 and, Lactobacillus acidophilus LA-5-containing yoghurt, on fecal bacterial counts of healthy adults. Int J Food Microbiol. 2011 Sep 1;149(1):50-7. doi: 10.1016/j.ijfoodmicro.2010.12.026. Epub 2011 Jan 15. PMID 21296446